CLINICAL TRIAL: NCT07331649
Title: Comparative Effects of Modified Tabata Training and Fartlek Training on Strength, Power and Endurance in Amateur Football Players
Brief Title: Comparative Effects of Modified Tabata Training and Fartlek Training in Amateur Football
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/24/0495
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Sports Physical Therapy
Keywords: Modified Tabata Training; Fartlek Training; Amateur Football Players

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Outcomes Assessor
Masking Description: The Outcome Assessors are Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 40 Participants will be in Group A. They will Perform Modified Tabata Training.
  Interventions: Other: Modified Tabata Training
- Group B (Active Comparator): 40 participant will be Group B. They will perform Fartlek Training.
  Interventions: Other: Fartlek Training

INTERVENTIONS:
Other: Modified Tabata Training — The Modified Tabata training Program that will be carried out for 3 sessions per week over 6 weeks is as follows: there will be 3 training sessions in a week. In first two weeks, the 24-minute session will be divided into 6 sets, each set lasting 4 minutes consist of 8 rounds, with a 2-minute rest period between each set. The 4 minute exercise duration will consist of a work-to-rest ratio of 20 seconds of work and 10 seconds of rest
  Arms: Group A
Other: Fartlek Training — fartlek session begins with a warm-up, followed by intervals of intense effort (e.g., 2, 3, 4, 3, 2 minute hard and moderate runs) with recovery periods (2 minutes) in between, then concludes with a cool-down.
  Arms: Group B

SUMMARY:
Background: Football requires players to excel in both high-intensity, fast-paced actions and slower moments of rest, which demand a range of well-developed motor skills, including power, endurance and strength. Endurance enables players to maintain prolonged physical effort without diminishing performance, a necessity given the sport's demand for players to cover 9-14 km per game, with up to 15% of this distance covered in high-intensity sprints. Strength is also crucial, helping players perform actions such as jumping, pushing during sprints, and maintaining stability, all of which enhance performance and resilience on the field. To adapt to the changing physical demands of football, training methods like treadmill sprint training and fartlek training (FT) are commonly used, each with different impacts on physiological development. Objective: The objective of this study is to compare the effects of treadmill sprint training and fartlek training on leg press strength, power and endurance on amateur football players. Methodology: A sample size of 42 football players will be randomly allocated to either fartlek training group or modified Tabata training group. A typical fartlek session begins with a warm-up, followed by intervals of intense effort (e.g., 2, 3, 4, 3, 2 minute hard and moderate runs) with recovery periods (2 minutes) in between, then concludes with a cool-down. This 2, 3, 4, 3, 2 interval set helps athletes improve endurance, strength and power and adapt to varied game-like conditions. The Modified Tabata training Program that will be carried out for 3 sessions per week over 6 weeks is as follows: there will be 3 training sessions in a week. In first two weeks, the 24-minute session will be divided into 6 sets, each set lasting 4 minutes consist of 8 rounds, with a 2-minute rest period between each set. The 4 minute exercise duration will consist of a work-to-rest ratio of 20 seconds of work and 10 seconds of rest. The level of exercise progressively increased throughout the 6-week program, by increasing the set of exercise Outcome measures in the both groups will be assessed by Squats test, Vertical jump test,3-min step up test and Yo-Yo Intermittent recovery test . All these measures will be taken at the baseline and again after 6 weeks of training to assess the effectiveness of the training program and the resulting improvements in strength, power, and endurance.

DETAILED DESCRIPTION:
Study design: Randomized clinical trial Sample size: calculated by Epitool is 40 (20 in each group) Sampling technique: Non-probability convenient sampling Study setting Al-Musaddiq Institute of Higher Education, Kharian FG Degree College for Boys, Kharian cantt.

Inclusion:

Young Male football player aged 18-25 years Amateur football players (who are in practice from last 8 months) Athletes with BMI 18.5kg/m2 -24.9kg/m2 The participants not taking any supplements or anabolic steroids Engages in other physical activities (e.g., gym, running) at least weekly. Exclusion The participants with history of a severe injury (e.g. ACL tear, fracture ) in the last 6 months History of any lower limb surgery (e.g., ACL reconstruction or any major surgery) Any musculoskeletal disorder. Chronic respiratory conditions (e.g., COPD, severe asthma) affecting exercise capacity. Significant weight fluctuations in the past 3 months. Any diagnosed psychological and cardiovascular conditions that could affect participation. Tools For strength: squats test (ICC=0.99) For power: Vertical jump test (ICC = 0.968) For endurance: 3-min step up test (ICC = 0.913) , Yo Yo intermittent recovery Test (ICC= between 0.87 and 0.95)

ELIGIBILITY:
Inclusion Criteria:

* Young Male football player aged 18-25 years.
* Amateur football players (who are in practice from last 8 months)
* Athletes with BMI 18.5kg/m2 -24.9kg/m2.
* Engages in other physical activities (e.g., gym, running) at least weekly.
* The participants not taking any supplements or steroids.

Exclusion Criteria:

* The participants with a history of a severe injury (e.g. ACL tear, fracture ) in the last 6 months.
* History of any lower limb surgery (e.g., ACL reconstruction or any major surgery)
* Any musculoskeletal disorder.
* Chronic respiratory conditions (e.g., COPD, severe asthma) affecting exercise capacity.
* Significant weight fluctuations in the past 3 months.
* Any diagnosed psychological and cardiovascular conditions that could affect participation.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-10-05 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Squat Test | 6 weeks
  The squats test was used to assess the strength of the lower limbs, clearly indicating the players' ability to generate force through their legs, which is crucial for movements such as sprinting and jumping in football.
Vertical Jump Test | 6 weeks
  The vertical jump test was utilized to measure explosive power, an essential component for effective performance in football, as it directly relates to a players ability to jump for headers or evade opponents.
3-minute step-up Test | 6 weeks
  To measure cardiovascular endurance, 3-minute step-up test was used, which evaluates the players' ability to sustain activity over time, reflecting their cardiovascular fitness and stamina on the field.
YoYo intermittent recovery Test | 6 weeks
  To Measure speed Endurance, YoYo intermittent recovery test was used, which evaluate the athlete´s speed endurance, aerobic capacity and fitness level. By completing YoYo intermittent recovery test, players demonstrate their ability to sustain intense physical activity, change direction quickly and maintain speed.

CONTACTS AND LOCATIONS:
Overall Officials: Afifa Tariq, Principal Investigator — Riphah International University
Locations (1):
- Al Mussadiq Institute of Higher Education, Kharian, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaouachi A, Brughelli M, Chamari K, Levin GT, Ben Abdelkrim N, Laurencelle L, Castagna C. Lower limb maximal dynamic strength and agility determinants in elite basketball players. J Strength Cond Res. 2009 Aug;23(5):1570-7. doi: 10.1519/JSC.0b013e3181a4e7f0. PMID 19620905
- [Background] Bret C, Rahmani A, Dufour AB, Messonnier L, Lacour JR. Leg strength and stiffness as ability factors in 100 m sprint running. J Sports Med Phys Fitness. 2002 Sep;42(3):274-81. PMID 12094115
- [Background] Hori N, Newton RU, Andrews WA, Kawamori N, McGuigan MR, Nosaka K. Does performance of hang power clean differentiate performance of jumping, sprinting, and changing of direction? J Strength Cond Res. 2008 Mar;22(2):412-8. doi: 10.1519/JSC.0b013e318166052b. PMID 18550955
- [Background] Nowak M, Szymanek-Pilarczyk M, Stolarczyk A, Oleksy L, Muracki J, Wasik J. Normative and limit values of speed, endurance and power tests results of young football players. Front Physiol. 2025 Jan 8;15:1502694. doi: 10.3389/fphys.2024.1502694. eCollection 2024. PMID 39844899
- [Background] Di Giminiani R, Visca C. Explosive strength and endurance adaptations in young elite soccer players during two soccer seasons. PLoS One. 2017 Feb 13;12(2):e0171734. doi: 10.1371/journal.pone.0171734. eCollection 2017. PMID 28192512
- [Background] Modric T, Versic S, Sekulic D. Position Specific Running Performances in Professional Football (Soccer): Influence of Different Tactical Formations. Sports (Basel). 2020 Dec 10;8(12):161. doi: 10.3390/sports8120161. PMID 33321874